CLINICAL TRIAL: NCT00548080
Title: A Non-Comparative, Multicenter, Open-Label, Study to Evaluate the Safety and Efficacy of Caspofungin Acetate as Empirical Therapy in Chinese Adults With Persistent Fever and Neutropenia
Brief Title: Evaluate the Safety and Efficacy of Caspofungin Acetate as Empirical Therapy in Chinese Adults With Persistent Fever and Neutropenia (0991-055)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0991-055; 2007_032
Record Dates: First submitted 2007-10-19; First posted 2007-10-23 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Fungal Infection
MeSH Terms: conditions — Mycoses | interventions — Caspofungin; Duration of Therapy

INTERVENTIONS:
Drug: MK0991, caspofungin acetate / Duration of Treatment:

SUMMARY:
Registration study

ELIGIBILITY:
Inclusion Criteria:

* Patient has had an absolute neutrophil count < 500/mm3 for at least 96 hours (the patient must not be expected to recover from neutropenia in the next 48 hours), and has received at least 96 hours of parenteral broad spectrum systemic antibacterial therapy preceding study entry, and patient has fever >38.0 Degrees Centigrade within the last 24 hours prior to study entry

  * Appropriate antibiotics are those that provide broad spectrum gram-positive and gram-negative coverage

Exclusion Criteria:

* Patient has an inadequately managed bacterial infection at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2006-03; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
The proportion of caspofungin-treated patients with SAE

SECONDARY OUTCOMES:
The proportion of caspofungin-treated patients with a favorable efficacy response at the end of caspofungin study therapy

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC